CLINICAL TRIAL: NCT06417580
Title: Effect of Experimental Pregabalin Gel in Controlling Cervical Dentin Hypersensitivity: a Randomized, Double-blind, Controlled Clinical Study
Brief Title: Effect of Pregabalin Gel in Controlling Cervical Dentin Hypersensitivity
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jesuína Lamartine Nogueira Araújo (Other)
Responsible Party: Sponsor-Investigator, Jesuína Lamartine Nogueira Araújo, Coordinator and professor of the Postgraduate Program in Dentistry at Universidade Federal do Pará, Universidade Federal do Para
Organization: Universidade Federal do Para (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ppgoufpa
Record Dates: First submitted 2024-04-11; First posted 2024-05-16 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Dentin Sensitivity
Keywords: pregabalin; dental sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: This randomized clinical trial will be parallel, double-blind, placebo-controlled. Composed of three groups: a placebo control group with gel without any active ingredient (CG), a group with potassium nitrate gel (GNK) and an experimental group with 10% potassium pregabalin gel (GPG). Applications will be carried out in 3 sessions with an interval of 72 hours between each one. Sensitivity recording will be performed at T0 (baseline), T1 (after first session), T2 (after second session), T3 (after third session), T4 (7 days after the last session) and T5 (one month after the last session) and T6 (3 months after the last session).
  A questionnaire (QEDH-15) will be applied to evaluate the impact of desensitizing treatment on improving the participants' oral health-related quality of life (HRQoL). The questionnaire will be applied at baseline (T0) and at the last sensitivity record (T6).
Who Masked: Participant, Investigator
Masking Description: This double-blind study guarantees the confidentiality of the interventions, since both the research participant and the main researcher will not be able to differentiate the procedure applied. The placebo gel, the experimental desensitizing gel and the potassium nitrate gel will be inserted into a dappen jar delivered immediately before the clinical interventions by a research collaborator. The gels have a similar texture, color and odor to prevent identification. The evaluator will also not be aware of the group the participant belonged to, as they will not participate in the randomization process. The research will have a single operator to carry out the clinical part.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Negative Control Group (Placebo Comparator): A negative control group with gel without any active ingredient.
  The protocol used for all groups will be the same: prophylaxis with an extra soft robinson brush and pumice stone, insertion of retractor thread number #000 in the gingival sulcus and then application and friction of the placebo gel with a microbrush applicator for 10 seconds, which will remain in contact with the tooth surface for 10 minutes, and the excess will be subsequently removed. Three desensitizing treatment sessions will be carried out, with an interval of 72 hours between each session.
  Interventions: Other: Placebo Treatment
- Positive Control Group (Active Comparator): Potassium nitrate gel group that will serve as a positive control
  The protocol used for all groups will be the same: prophylaxis with an extra soft robinson brush and pumice stone, insertion of retractor thread number #000 in the gingival sulcus and then application and friction of the potassium nitrate gel with a microbrush applicator for 10 seconds, which will remain in contact with the tooth surface for 10 minutes, and the excess will be subsequently removed. Three desensitizing treatment sessions will be carried out, with an interval of 72 hours between each session.
  Interventions: Other: Nitrate Potassium Treatment
- Experimental group (Experimental): Experimental group with 10% pregabalin gel.
  The protocol used for all groups will be the same: prophylaxis with an extra soft robinson brush and pumice stone, insertion of retractor thread number #000 in the gingival sulcus and then application and friction of the pregabalin gel with a microbrush applicator for 10 seconds, which will remain in contact with the tooth surface for 10 minutes, and the excess will be subsequently removed. Three desensitizing treatment sessions will be carried out, with an interval of 72 hours between each session.
  Interventions: Other: Pregabalin Treatment

INTERVENTIONS:
Other: Placebo Treatment — Desensitizing protocol with none active ingredient to evaluate the control of cervical dentin hypersensitivity
  Arms: Negative Control Group
Other: Nitrate Potassium Treatment — Desensitizing protocol with potassium nitrate gel to analyze and compare with other groups the effects of controlling cervical dentin hypersensitivity
  Arms: Positive Control Group
Other: Pregabalin Treatment — Desensitizing protocol with experimental 10% pregabalin gel to evaluate the control of cervical dentin hypersensitivity
  Arms: Experimental group

SUMMARY:
This randomized, double-blind, placebo-controlled clinical study aims to evaluate the effect of a gel formulation based on 10% of pregabalin in the treatment of HD and on the participants' quality of life. The sample calculation will be based on previous work. After selecting participants, the participants will be randomly assigned to the following groups: placebo control group (CG), potassium nitrate gel group (GNK) and pregabalin gel group (GPG). A questionnaire (QEDH-15) to assess the impact of desensitizing treatment on oral health-related quality of life (OHRQoL) will be applied at baseline (T0) and in the last sensitivity record (T6). Pain will be assessed using a visual analogue scale after evaporative stimulation with an air jet and tactile stimulation with an exploratory probe. Three desensitizing treatment sessions will be carried out, with an interval of 72 hours between them. Sensitivity recording will be performed at T0 (baseline), T1 (after the first session), T2 (after the second session), T3 (after the third session), T4 (7 days after the last session), T5 (one month after the last session) and T6 (3 months after the last session). Data will be collected and subjected to statistical analysis for parametric data (ANOVA followed by Student-Newman-Keuls) or non-parametric data (Friedman's ANOVA followed by Tukey). To analyze the impact on quality of life, the Friedman test will be used.

DETAILED DESCRIPTION:
To obtain the experimental pregabalin gel, a carbopol 940 gel base was used. To prepare the base gel for the formulation, each component was weighed on an analytical balance and, after 24 hours, the components were taken to a mechanical shaker, rotating at 1000 rpm for 10 minutes. 50% triethanolamine was added to adjust the pH to ±6 and complete gel formation. The concentrations of the components of the initial base formula were adjusted to obtain a homogeneous, transparent gel with good consistency. A PG solution (10 mg/ml) was prepared by diluting the drug, which is presented as a white, crystalline powder (Vardhman Chemtech Ltd, Punjab, India), with purified water. The solution was stirred for 10 min in a water bath (Taitec) and centrifuged at 4°C for 10 min. The supernatant obtained was collected and then incorporated into the 1% carbopol-based gel.

This formulation has already been evaluated in a previous study regarding quality standards, physical/chemical characterization, cytotoxicity and subjected to stability analyzes (preliminary and accelerated). Its characteristics indicate that it is a favorable formulation for clinical application.

This randomized clinical study will follow the guidelines for clinical trials recommended by CONSORT (Consolidated Standards Of Reporting Trials) and will be submitted to the Human Research Ethics Committee of the Institute of Health Sciences at the Federal University of Pará (CEP-ICS/UFPA). All selected participants who agree to participate in the research will be informed about the benefits, risks, methods, and goals of the study before consenting to their participation through the Informed Consent Form declaring that the participants agree with all the steps to be taken. The participants can withdraw from the research at any time, following the principles of the Declaration of Helsinki.

This randomized clinical trial will be parallel, double-blind, placebo-controlled and all clinical interventions will be conducted in the clinics of the Faculty of Dentistry of the Federal University of Pará (FOUFPa). The research will consist of three groups: a placebo control group (CG) with gel without any active ingredient, a group with potassium nitrate gel (Ultradent, South Jordan, UT, USA) (GNK), and an experimental group with gel 10% Pregabalin (GPG). Applications will be carried out in 3 sessions with an interval of 72 hours between each one. Sensitivity recording will be performed at T0 (baseline), T1 (after the first session), T2 (after the second session), T3 (after the third session), T4 (7 days after the last session), and T5 (one month after the last session) and T6 (3 months after the last session).

A questionnaire (QEDH-15) will be applied to evaluate the impact of desensitizing treatment on improving the participants' oral health-related quality of life (HRQoL). The questionnaire will be applied at baseline (T0) and the last sensitivity record (T6). Higher QEHD-15 scores indicate a negative impact on the oral health-related quality of life (OHRQoL) of research participants.

The sample size was determined using the GPower 3.1 program (Heinrich-Heine-Universität Düsseldorf, Germany), based on a comparison of intergroup means. According to previous studies, the minimum expected difference is 2.26, and a standard deviation of 2 between groups. An alpha of 5%, power of 80%, and a 20% increase in possible loss of participants were considered. The final sample size determined was 63 teeth in total, 21 sensitive teeth per group.

To evaluate the painful sensation of hypersensitivity, a Visual Analogue Scale (VAS) will be used. The initial mark "0" represents no pain and the opposite mark "10" represents extreme pain.

The participant will be asked to signal the number compatible with the painful sensation after applying the evaporative stimulus, by applying a jet of air from a triple syringe for two seconds, at room temperature, perpendicular to the buccal surface of the tooth at a distance of 1cm, and also by tactile stimulation, where a cross-shaped exploring probe will slide into the cervical region of the hypersensitive teeth, vertically in the cervical-incisal direction and horizontally in the mesiodistal direction. These stimuli will be performed after relative individual isolation with isolation tape (Isotape, Septodont, Louisville, USA) and cotton rolls (Dental Cremer, SC, Brazil).

Random distribution between the groups will be carried out in a block, through a numerical draw that allows each participant to be allocated into one of the three groups (GC, GNK and GPG) using Biostat 5.3 software (Instituto Mamirauá, PA, Brazil). The confidentiality of the allocation will be maintained throughout the sample formation process, through a numerical draw with numbered and coded papers. All participants and the clinical operator will not know the group's codes.

This double-blind study guarantees the confidentiality of the interventions since both the research participant and the main researcher will not be able to differentiate the procedure applied. The placebo gel, the experimental desensitizing gel, and the potassium nitrate gel will be inserted into a dappen jar and delivered immediately before the clinical interventions by a research collaborator. The gels have a similar texture, color and odor to prevent identification. The evaluator will also not be aware of the group the participant belonged to, as the clinical operator will not participate in the randomization process. The research will have a single operator to carry out the clinical part.

The data will be analyzed for normality of distribution, using the Shapiro-Wilk test. If it presents a normal distribution, the ANOVA parametric analysis will be used to verify the existence of differences between the group means and the Student-Newman-Keuls post-hoc test will be used to verify the differences between the times. In case of abnormal distribution, the Friedman repeated measures test and the Tukey post hoc test will be used. To analyze differences in quality of life-related to oral health at T0 and T6, the Friedman test will be used. Data analysis will be performed using the freely available statistical software Jamovi (Version 2.3). The significance level α will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Sensitive teeth with a response ≥ 04 on the visual analog scale (VAS) to tactile and evaporative stimuli;
* Dentin exposure in anterior and/or posterior teeth, either due to the presence of non-carious cervical lesions and/or gingival recession.

Exclusion Criteria:

* Allergic to the active ingredient and/or components of the formulation;
* Carious lesions and/or dental pulpitis;
* Recent medication with analgesics or anti-inflammatories;
* Received desensitizing treatment, orthodontic treatment, or having undergone tooth whitening up to six months prior baseline.
* Large restorations in sensitive teeth
* Eating disorders (bulimia, anorexia,...)
* Periodontal disease (moderate to severe)
* Bruxism
* Cracks or fractures in the enamel;
* Pregnant or breastfeeding women.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-05-28 (Estimated); Primary Completion 2024-09-28 (Estimated); Study Completion 2024-09-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with dentin hypersensitivity: an average of 6 participants and 21 sensitive teeth in the group. | Through study completion, an average of 3 months for each participant
  The use of 10% pregabalin gel influence in the painful symptoms of dentin hypersensitivity. The results will be evaluated through study completion, an average of 3 months for each participant. The data will tell if the positive results were of short, medium and long-term.

CONTACTS AND LOCATIONS:
Overall Officials: Jesuina L Nogueira Araujo, Doctor, Principal Investigator — Federal University of Pará

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Barros APO, de Melo Alencar C, de Melo Pingarilho Carneiro A, da Silva Pompeu D, Barbosa GM, Araujo JLN, Silva CM. Combination of two desensitizing protocols to control dentin hypersensitivity in non-carious lesions: a randomized, double-blind clinical trial. Clin Oral Investig. 2022 Feb;26(2):1299-1307. doi: 10.1007/s00784-021-04104-2. Epub 2021 Aug 5. PMID 34351504
- [Background] Douglas-De-Oliveira DW, Lages FS, Paiva SM, Cromley JG, Robinson PG, Cota LOM. Cross-cultural adaptation of the Brazilian version of the Dentine Hypersensitivity Experience Questionnaire (DHEQ-15). Braz Oral Res. 2018;32:e37. doi: 10.1590/1807-3107bor-2018.vol32.0037. Epub 2018 May 3. PMID 29723336
- [Background] Tolentino AB, Zeola LF, Fernandes MRU, Pannuti CM, Soares PV, Aranha ACC. Photobiomodulation therapy and 3% potassium nitrate gel as treatment of cervical dentin hypersensitivity: a randomized clinical trial. Clin Oral Investig. 2022 Dec;26(12):6985-6993. doi: 10.1007/s00784-022-04652-1. Epub 2022 Jul 25. PMID 35871702
- [Background] Sgreccia PC, Dame-Teixeira N, Barbosa RES, Araujo PF, Zanatta RF, Garcia FCP. Assessment of the Oral Health Impact Profile (OHIP-14) improvement of different treatments for dentin hypersensitivity in noncarious cervical lesions-a randomized clinical study. Clin Oral Investig. 2022 Nov;26(11):6583-6591. doi: 10.1007/s00784-022-04610-x. Epub 2022 Jul 7. PMID 35796800